CLINICAL TRIAL: NCT04525326
Title: A Prospective Study on the Conversion Therapy of Ras / BRAF Wild Type Right-sided Colon Cancer Patients With Initially Unresectable Liver Metastases: Standard Chemotherapy Plus Cetuximab VS. Standard Chemotherapy Plus Bevacizumab
Brief Title: Conversion Therapy of RAS/BRAF Wild-Type Right-sided Colon Cancer Patients With Initially Unresectable Liver Metastases
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHENKANG2020XU
Record Dates: First submitted 2020-08-21; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Colorectal Cancer; Liver Metastases
Keywords: Cetuximab; Bevacizumab; Liver Metastases; Colorectal Cancer; right-sided
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard chemotherapy plus Cetuximab (Experimental)
  Interventions: Drug: Cetuximab; Drug: mFOLFOX/FOLFIRI ( Standard Chemotherapy)
- standard chemotherapy plus Bevacizumab (Experimental)
  Interventions: Drug: Bevacizumab; Drug: mFOLFOX/FOLFIRI ( Standard Chemotherapy)

INTERVENTIONS:
Drug: Cetuximab — mFOLFOX+Cetuximab for Ras / BRAF Wild Type Unresectable Right Colon Cancer Patients With Liver Metastasis
  Arms: standard chemotherapy plus Cetuximab
Drug: Bevacizumab — mFOLFOX+Bevacizumab for Ras / BRAF Wild Type Unresectable Right Colon Cancer Patients With Liver Metastasis
  Arms: standard chemotherapy plus Bevacizumab
Drug: mFOLFOX/FOLFIRI ( Standard Chemotherapy) — Standard Chemotherapy

SUMMARY:
The prognosis of patients with metastatic right-sided colon cancer is worse than that of patients with metastatic left-sided cancer. Different guidelines have different recommendations on specific conversion therapy for colorectal liver metastases. The United States NCCN guidelines do not recommend standard chemotherapy combined with anti EGFR monoclonal antibody for patients with right colon cancer. The European ESMO guidelines recommend that patients with Ras / BRAF wild-type right-sided colon cancer should first consider three drugs ± bevacizumab, but considering the objective response rate results, standard chemotherapy + anti EGFR monoclonal antibody is still one of the choices. China CSCO guidelines recommend standard chemotherapy ± bevacizumab, and also recommend standard chemotherapy + cetuximab for patients with right-sided colon cancer.

Therefore, the targeted therapy for RAS / BRAF wild-type metastatic right colon cancer is still controversial. Therefore, we are ready to carry out the clinical trial of cetuximab and bevacizumab in conversion therapy for RAS / BRAF wild-type metastatic right colon cancer. The conversion resection rate is the primary point, and the objective response rate, perioperative safety and long-term survival are the secondary points.

ELIGIBILITY:
Inclusion Criteria:

1. The primary tumor was confirmed by histology as colorectal adenocarcinoma
2. primary right-sided colorectal adenocarcinoma
3. Radiologic evidence suggests that the initial unresectable liver metastases
4. RAS/BRAF gene wild-type states
5. ECOG was 0 ~ 1
6. Life expectancy ≥ 3 months
7. Good hematological function: neutrophil ≥ 1.5x109/l and platelet count ≥ 100x109 / L; HB ≥ 9g / dl (within one week before randomization)
8. Normal liver and kidney function: serum bilirubin ≤ 1.5x normal upper limit (ULN), alkaline phosphatase ≤ 5x ULN, serum transaminase (AST or ALT) ≤ 5x ULN (within one week before randomization);
9. Sign the written informed consent to participate in the experiment

Exclusion Criteria:

1. Patients with liver metastases from colorectal cancer who have previously received targeted therapy, chemotherapy, radiotherapy or interventional therapy
2. Known or suspected extrahepatic metastasis
3. Patients with known hypersensitivity to any component of the study treatment
4. Clinical related coronary heart disease or history of myocardial infarction in the last 12 months or left ventricular ejection fraction below normal range
5. Acute or subacute intestinal obstruction
6. Pregnancy (no pregnancy confirmed by serum / urine β - hCG) or breastfeeding.
7. She had other malignant tumors within 5 years, except for those with skin basal cell carcinoma or cervical cancer
8. Known drug / alcohol abuse
9. No legal capacity or limited legal capacity
10. There is peripheral neuropathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Conversion liver resection rate | up to 6 months
  Rate of conversion from initially unresectable liver metastases to resectable ones

SECONDARY OUTCOMES:
objective response rate | up to 6 months
  rate of objective response for therapy(according to RECIST 1.0)
Incidence of adverse events | up to 6 months
  Incidence of adverse events
Progression free survival | up to 3 years
  Progression free survival
overall survival | up to 5 years
  overall survival

IPD SHARING:
Plan to Share IPD: No